CLINICAL TRIAL: NCT02034500
Title: A Phase 1, Randomized, Placebo Controlled, Single Center, Dose Escalation Study to Evaluate the Safety and Immunogenicity of 3 Vaccinations With Shigella Sonnei Vaccine (1790GAHB) Administered Either by Intradermal, Intranasal or Intramuscular Route in Healthy Adults.
Brief Title: Evaluate a New Shigella Sonnei Vaccine Administered Either by Intradermal, Intranasal or Intramuscular Route in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GSK Vaccines Institute For Global Health S.r.l. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: H03_02TP
Record Dates: First submitted 2014-01-02; First posted 2014-01-13 (Estimated); Last update posted 2016-06-21 (Estimated); Status verified 2016-06

CONDITIONS: Shigellosis
Keywords: prevention; Shigella sonnei
MeSH Terms: conditions — Dysentery, Bacillary

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (10):
- S. sonnei 1790GAHB - 0.1 mcg - ID (Experimental): Subjects enrolled in COHORT A receiving 3 injections of S. sonnei 1790GAHB - 0.1 mcg intradermally (ID)
  Interventions: Biological: S. sonnei 1790GAHB
- S. sonnei 1790GAHB - 1 mcg - ID (Experimental): Subjects enrolled in COHORT B receiving 3 injections of S. sonnei 1790GAHB - 1 mcg intradermally (ID)
  Interventions: Biological: S. sonnei 1790GAHB
- S. sonnei 1790GAHB - 10 mcg - ID (Experimental): Subjects enrolled in COHORT C receiving 3 injections of S. sonnei 1790GAHB - 10 mcg intradermally (ID)
  Interventions: Biological: S. sonnei 1790GAHB
- S. sonnei 1790GAHB - 5 mcg - IN (Experimental): Subjects enrolled in COHORT A receiving 3 injections of S. sonnei 1790GAHB - 5 mcg intranasally (IN)
  Interventions: Biological: S. sonnei 1790GAHB
- S. sonnei 1790GAHB - 20 mcg - IN (Experimental): Subjects enrolled in COHORT B receiving 3 injections of S. sonnei 1790GAHB - 20 mcg intranasally (IN)
  Interventions: Biological: S. sonnei 1790GAHB
- S. sonnei 1790GAHB - 80 mcg - IN (Experimental): Subjects enrolled in COHORT C receiving 3 injections of S. sonnei 1790GAHB - 80 mcg intranasally (IN)
  Interventions: Biological: S. sonnei 1790GAHB
- S. sonnei 1790GAHB - 5 mcg - IM (Experimental): Subjects enrolled in COHORT C receiving 3 injections of S. sonnei 1790GAHB - 5 mcg intramuscularly (IM)
  Interventions: Biological: S. sonnei 1790GAHB
- Placebo - ID (Placebo Comparator): 2 subjects enrolled in each COHORT A, B and C receiving 3 injections of Placebo intradermally (ID). These were pooled in one Placebo group in the analyses
  Interventions: Biological: Placebo
- Placebo - IN (Placebo Comparator): 2 subjects enrolled in each COHORT A, B and C receiving 3 injections of Placebo intranasally (IN). These were pooled in one Placebo group in the analyses
  Interventions: Biological: Placebo
- Placebo - IM (Placebo Comparator): 2 subjects enrolled in COHORT C receiving 3 injections of Placebo intramuscularly (IM)
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: S. sonnei 1790GAHB
  Other Names: Shigella sonnei vaccine
  Arms: S. sonnei 1790GAHB - 0.1 mcg - ID; S. sonnei 1790GAHB - 1 mcg - ID; S. sonnei 1790GAHB - 10 mcg - ID; S. sonnei 1790GAHB - 20 mcg - IN; S. sonnei 1790GAHB - 5 mcg - IM; S. sonnei 1790GAHB - 5 mcg - IN; S. sonnei 1790GAHB - 80 mcg - IN
Biological: Placebo
  Arms: Placebo - ID; Placebo - IM; Placebo - IN

SUMMARY:
This Phase 1 clinical trial is aimed to evaluate the safety and immunogenicity of 3 doses of a candidate vaccine against Shigella sonnei (1790GAHB vaccine) when administered at different dosages by different routes (intradermally, intranasally or intramuscularly) in healthy adults (18 to 45 years of age at enrollment). The safety profile of the 1790GAHB vaccine is evaluated in comparison to that of placebo (GAHB-Placebo), constituted by an aluminum hydroxide suspension having the same concentration as study vaccine formulations. A total of 52 eligible subjects will be assigned to one of three sequential cohorts as follows:

Cohort A) 0.1 μg ID and 5 μg IN Cohort B) 1 μg ID and 20 μg IN Cohort C) 10 μg ID, 80 μg IN and 5 μg IM Within each cohort, in an observer-blind fashion, subjects will be randomized to receive three vaccinations, four weeks apart, of either 1790GAHB vaccine (at five antigen concentrations) or GAHB placebo. Specifically for IN and ID administration routes, a Data Safety Monitoring Board will be in place to receive a summary of all safety data obtained during one week follow-up post-first vaccination with the lower dose. Based on evaluation of the safety data, the Data Safety Monitoring Board will make a recommendation, as to whether the next cohort should be vaccinated with higher antigen concentration or not.

Expected duration of the study for an individual subject is 9 months. Each subject will be followed-up for 6 months after the 3rd vaccination

ELIGIBILITY:
Inclusion Criteria:

1. Males and females of age ≥18 years to ≤45 years.
2. Individuals who, after the nature of the study have been explained to them, have given written consent according to local regulatory requirements.
3. Individuals in good health as determined by the outcome of medical history, physical examination, hematology, renal, bone and liver panels (including negative for agglutination testing of S. sonnei), urinalysis and clinical judgment of the investigator.
4. If women of childbearing potential, have a negative pregnancy test prior to study vaccination and willingness to use acceptable contraceptive measures for the entire study duration.
5. Individuals available for follow-up for the duration of the study.
6. Individuals registered with a general practitioner.

Exclusion Criteria:

1. Individuals with a history of recurrent wheezing, asthma, respiratory allergies, allergic rhinitis, nasal surgery or significant nasal abnormalities (e.g. polyps), and Bell's palsy. Presence of nasal piercings. Symptoms of upper respiratory tract infection within 3 days of intended study vaccination is a temporary exclusion criterion.
2. Individuals unwilling to abstain from medications or other agents that are applied via the nasal route from 24 hours prior to each nasal dosing through to the safety assessment 1 week later.
3. Individuals with behavioral or cognitive impairment or psychiatric disease that, in the opinion of the investigator, may interfere with the subject's ability to participate in the study.
4. Individuals with any progressive or severe neurological disorder, seizure disorder or Guillain-Barré syndrome.
5. Individuals who are not able to understand and to follow all required study procedures for the whole period of the study.
6. Individuals with history of any illness that, in the opinion of the investigator, might interfere with the results of the study or pose additional risk to the subjects due to participation in the study.
7. Individuals with human leukocyte antigen (HLA) -B27 positive and/or with history of reactive arthritis
8. Individuals with known HIV, HBV and HCV infection or HIV related disease, with history of an autoimmune disorder or any other known or suspected impairment /alteration of the immune system, or under immunosuppressive therapy including use of systemic corticosteroids or chronic use of inhaled high-potency corticosteroids within the previous 30 days, or were in chemotherapy treatment within the past 6 months.
9. Individuals with a known bleeding diathesis, or any condition that may be associated with a prolonged bleeding time.
10. Individuals with any serious chronic or progressive disease according to judgment of the investigator (e.g., neoplasm, insulin dependent diabetes, cardiac, renal or hepatic disease).
11. Individuals who have any malignancy or lymphoproliferative disorder.
12. Individuals with history of allergy to vaccine components.
13. Individuals participating in any clinical trial with another investigational product 90 days prior to first study visit or intent to participate in another clinical study at any time during the conduct of this study.
14. Individuals who received any other vaccines within 4 weeks prior to enrollment in this study or who are planning to receive any vaccine within the entire study duration except influenza vaccination, which is not allowed within the period included between 4 weeks before 1st vaccination and 4 weeks after 3rd vaccination
15. Individuals who have received blood, blood products and/or plasma derivatives including parenteral immunoglobulin preparations in the past 12 weeks.
16. Individuals who are part of study personnel or close family members to the personnel conducting this study or employees of the clinical trial site institution.
17. Individuals with body temperature > 38.0 degrees Celsius within 3 days of intended study vaccination.
18. BMI > 30 kg/m2.
19. Individuals with history of substance or alcohol abuse within the past 2 years.
20. Women who are pregnant or breast-feeding or of childbearing age who have not used or do not plan to use acceptable birth control measures, for the duration of the study.
21. Females with history of stillbirth, neonatal loss, or previous infant with anomaly.
22. Individuals who have a previously ascertained or suspected disease caused by S. sonnei or positive S. sonnei serology at screening
23. Individuals who have had household contact with/and or intimate exposure to an individual with laboratory confirmed S. sonnei
24. Any condition, which, in the opinion of the investigator may pose an increased and unreasonable safety risk to the subject if participating to the present study

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2014-03; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Number of subjects with solicited local reaction after any vaccination | During a 7-day (Days 1-7) post vaccination period following any injection
  Any erythema/induration/swelling refers to: ≥25 mm in diameter. Grade 3 (severe) refers to erythema/induration/swelling >100 mm in diameter.
  Grade 3 (severe) for injection site pain/nasal pain/facial edema/rhinorrhea refers to: prevents daily activity
Number of subjects with solicited systemic reaction after any vaccination | During a 7-day (Days 1 to 7) post vaccination period following any injection
  Any= Incidence of any symptom regardless of intensity grade. Grade 3 = symptom that prevented daily activities
Number of subjects with Neutrophils results below and above the normal ranges | At Day 8
  Day 8: VISIT 2 (D7 post 1st vac)
Number of subjects with Neutrophils results below and above the normal | At Day 36
  Day 36: VISIT 3.1 (D7 post 2nd vac)
Number of subjects with Neutrophils results below and above the normal | At Day 57
  Day 57: VISIT 4 (3rd vac.)
Number of subjects with Neutrophils results below and above the normal | At Day 64
  Day 64: VISIT 4.1 (D7 post 3rd vac.)
Number of subjects with Neutrophils results below and above the normal | At Day 85
  Day 85: VISIT 5 (1 month post 3rd vac.)
Number of subjects with Neutrophils results below and above the normal | At Day 225
  Day 225: VISIT 6 (6 months post 3rd vac.)

SECONDARY OUTCOMES:
Anti-LPS S. sonnei serum IgG Geometric mean concentration (GMCs) | At baseline, at 28 days after each vaccination and at 168 days after last vaccination
Number of subjects with seroresponse for anti-LPS S. sonnei | At 28 days after each vaccination and 168 days after last vaccination
  Seroresponse is defined as: If half of the baseline value is greater than 25 ELISA Unit (EU) then an increase of at least 50% in the post-vaccination sample as compared to baseline [i.e. ((Post-vac minus baseline)/baseline)100% ≥ 50%]. If half of the baseline value is less or equal to 25 EU then an increase of at least 25 EU in the post-vaccination sample as compared to baseline (i.e. [post-vac minus baseline] ≥25 EU)
Number of subjects with high seroresponse for anti-LPS S. sonnei (IgG ELISA ≥121 EU) | At baseline, at 28 days after each vaccination and at 168 days after last vaccination
  High seroresponse is defined as a post vaccination titer ≥X anti-LPS serum IgG units in the GSK (former Novartis) ELISA that correspond to a titer of 1:800 in the ELISA method used by Cohen et al. (1989 J. Clin. Microbiol. 27:162). To determine the value for 'X' the GSK (former Novartis) anti-LPS ELISA was calibrated against the Cohen ELISA and it was found that a concentration of 121 EU EU/mL corresponds to a titer of 1:800 in the Cohen assay

CONTACTS AND LOCATIONS:
Overall Officials: David JM Lewis, MD, Principal Investigator — University of Surrey, Guildford, GU2 7XP United Kingdom
Locations (1):
- Surrey Clinical Research Center (Surrey CRC), Guildford, Surrey, United Kingdom

REFERENCES:
- [Derived] Launay O, Lewis DJM, Anemona A, Loulergue P, Leahy J, Scire AS, Maugard A, Marchetti E, Zancan S, Huo Z, Rondini S, Marhaba R, Finco O, Martin LB, Auerbach J, Cohen D, Saul A, Gerke C, Podda A. Safety Profile and Immunologic Responses of a Novel Vaccine Against Shigella sonnei Administered Intramuscularly, Intradermally and Intranasally: Results From Two Parallel Randomized Phase 1 Clinical Studies in Healthy Adult Volunteers in Europe. EBioMedicine. 2017 Aug;22:164-172. doi: 10.1016/j.ebiom.2017.07.013. Epub 2017 Jul 15. PMID 28735965
- [Derived] Muturi-Kioi V, Lewis D, Launay O, Leroux-Roels G, Anemona A, Loulergue P, Bodinham CL, Aerssens A, Groth N, Saul A, Podda A. Neutropenia as an Adverse Event following Vaccination: Results from Randomized Clinical Trials in Healthy Adults and Systematic Review. PLoS One. 2016 Aug 4;11(8):e0157385. doi: 10.1371/journal.pone.0157385. eCollection 2016. PMID 27490698